CLINICAL TRIAL: NCT07340125
Title: Effects of Pistachio Snacking on Metabolic Flexibility in Healthy Overweight and Obese Adults
Brief Title: Pistachio Snacking and Metabolic Flexibility
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Carolina (Other)
Collaborators: American Pistachio Growers (Other)
Responsible Party: Principal Investigator, Katie Hirsch, Assistant Professor, University of South Carolina
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Pro00145186
Record Dates: First submitted 2025-12-17; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Overweight (BMI > 25); Obese But Otherwise Healthy Participants; Overweight or Obese; Obese Patients (BMI ≥ 30 kg/m²); Poor Sleep Quality; Healthy Participants; Physically Inactive
Keywords: Pistachio; Tree Nuts; metabolic flexibility; metabolism; diet quality; snacking
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Intervention Model Description: Randomized, crossover
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pistachio (Experimental): Four days of pistachio snacking, to be consumed mid-morning (1oz; 9-11am), mid-afternoon (1oz; 2-4pm), and pre-sleep (0.5 oz; within 1hr of bedtime), while otherwise maintaining normal dietary habits. An addition snack will be consumed post-exercise (0.5oz).
  Interventions: Other: Pistachio
- Control (No Intervention): Maintain normal dietary habits for four days.

INTERVENTIONS:
Other: Pistachio — Roasted, lightly salted, pistachio kernels (no shell)
  Arms: Pistachio

SUMMARY:
The purpose of this study is to evaluate the effects of pistachio snacking on metabolic flexibility (at rest, during exercise, and in post-exercise recovery) in healthy overweight and obese adults. Secondary goals include evaluating effects on changes in diet quality, sleep characteristics, physical activity, and hormonal health in women. In randomized order, participants will complete four days of pistachio snacking and four days of normal dietary habits (control). For both conditions, primary outcomes of resting substrate metabolism, metabolic flexibility during exercise, and post-exercise substrate metabolism will be measured pre-post intervention via indirect calorimetry. Secondary outcome of diet quality (kcal, carb, fat, protein) will be measured pre-post intervention via diet log. Exploratory outcomes of daily physical activity (steps, intensity), nightly sleep characteristics (quantity, quality, latency, efficiency), and daytime sleepiness and hunger.

ELIGIBILITY:
Inclusion Criteria:

* Males and Females
* Age: 25-45 years
* Overweight or obese (BMI=25.0-34.9 kg/m²)
* Poor sleep quality (Pittsburgh Sleep Quality Index ≥ 5)
* Healthy (no diagnosed metabolic, cardiovascular, sleep, or other health condition that may significantly alter metabolism, sleep, or ability to participate in the exercise test)
* Not meeting weekly physical activity recommendations (<150 min moderate-intensity exercise, <75 minutes of vigorous-intensity exercise, and <2 days of strength training)
* Not following a diet that is restrictive or eliminates certain food group/types

Exclusion Criteria:

* Allergies to nuts, especially tree nuts
* Has a pacemaker
* Following a diet that is restrictive or eliminates certain food group/types
* Self-repoted health or disease state that may influence study outcomes, including known metabolic or endocrine disorder (e.g. prediabetes, type 1 or type 2 diabetes, or polycystic ovary syndrome), cardiovascular diseases, neuromuscular disorders, musculoskeletal disorders; current or recent history of cancer/cancer treatment (within the past year)
* History of gastrointestinal surgery, hysterectomy
* For women: pregnant or thinking of becoming pregnant during the time of participation, pregnant within the last year, currently breastfeeding, or known to be perimenopausal

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
resting metabolism | Day 0 and Day 5
  resting metabolic rate (RMR) and substrate utilization (RER) via indirect calorimetry
exercise metabolic flexibility | Day 0 and Day 5
  substrate metabolism (RER; indirect calorimetry) throughout a submaximal, graded exercise test
post-exercise metabolism | Day 0 and Day 5
  Energy expenditure and substrate metabolism (RER) measured at 0, 30, 60, 90min post-exercise via indirect calorimetry

SECONDARY OUTCOMES:
Caloric Intake | Day 0 and Day 4
  Average calorie intake (kcal) via 24-hr diet record
Carbohydrate Intake | Day 0 and Day 4
  Average carbohydrate intake (grams) via 24-hr diet record
Protein Intake | Day 0 and Day 4
  Average protein intake (grams) via 24-hr diet record
Fat Intake | Day 0 and Day 4
  Average fat intake (grams) via 24-hr diet record

OTHER OUTCOMES:
Physical Activity | daily continuous (Day 0 to Day 5)
  Daily (24-hr) steps and intensity minutes via wrist activity tracker
Sleep Quantity | Nightly (Day 0 to Day 5)
  Nightly sleep quantity (total time spent asleep; minutes) via wrist worn activity tracker.
Sleep Quality | Nightly (Day 0 to Day 5)
  Nightly sleep quality (time spent in deep sleep (minutes), REM sleep (minutes), and light sleep (minutes)) via wrist worn activity tracker.
Daytime sleepiness | Day 0 and Day 5
  Subjective likelihood of falling asleep in various situations via Epworth Sleepiness Scale. In this eight question survey, questions are rated on a scale of 0 (very unlikely) to 3 (very likely), with a total score of 0-9 indicating low daytime sleepiness, 10-15 indicating moderate daytime sleepiness, and 16-24 indicating severe daytime sleepiness.
Subjective hunger | Daily (Day 1 to Day 4)
  Degree of hunger/fullness (Visual Analog Scale) mid-morning (post-snack), late morning (a few hours post snack), and mid-afternoon (pre-snack).

CONTACTS AND LOCATIONS:
Overall Officials: Katie R Hirsch, PhD, Principal Investigator — University of South Carolina
Locations (1):
- Public Health Research Center: Clinical Exercise Research Center, Columbia, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No
data may be shared upon reasonable request.